CLINICAL TRIAL: NCT02420301
Title: Effects of Self-administered Exercises Based on Tuina Techniques on Musculoskeletal Disorders of Professional Orchestra Musicians
Brief Title: Effect of Self-administered Exercises on PRMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Cláudia Maria Gomes de Sousa, PhD student, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: claudiasousa_2
Record Dates: First submitted 2015-03-30; First posted 2015-04-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercises on real points (Experimental): Self administered exercises were done in real treatment points
  Interventions: Other: Tuina exercises
- Exercises on false points (Placebo Comparator): Self administered exercises were done in false treatment points
  Interventions: Other: Placebo Tuina exercises

INTERVENTIONS:
Other: Tuina exercises
  Arms: Exercises on real points
Other: Placebo Tuina exercises
  Arms: Exercises on false points

SUMMARY:
Objective: To study the effects of self-administered exercises based on tuina techniques on the pain intensity caused by playing related musculoskeletal disorders (PRMD) of professional orchestra musicians, using numeric visual scale (NVS).

Method: The investigators performed a prospective, controlled, single-blinded, randomized study with musicians suffering from PRMD. n= 69 musicians were randomly distributed into the experimental and into the control group. After an individual diagnostic assessment, specific tuina self-administered exercises were developed and taught to the participants. Musicians were instructed (educated) to repeat the exercises every day during 3 weeks. Pain intensity was measured by NVS before the intervention and after the 1st, 3rd, 5th, 10th, 15th and 20th days of self-exercising. The procedure was the same for the control group, however the Tuina exercises were executed in non-acupuncture points

ELIGIBILITY:
Inclusion Criteria:

* Professional orchestra musician presenting playing related musculoskeletal pain during at least 3 weeks

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Verbal numeric scale | At the baseline
Verbal numeric scale | After one day
Verbal numeric scale | After 3 days
Verbal numeric scale | After 5 days
Verbal numeric scale | After 10 days
Verbal numeric scale | After 15 days
Verbal numeric scale | After 20 days